CLINICAL TRIAL: NCT04759885
Title: Efficacy and Safety of mAnniTol in Bowel Preparation: Assessment of Adequacy and Presence of Intestinal levelS of Hydrogen and Methane During Elective Colonoscopy aFter mAnnitol or Standard Split 2-liter Polyethylene Glycol Solution Plus asCorbaTe - a Phase II/III, International, Multicentre, Randomized, Parallel-group, endoscOpist-bliNded, Dose-finding/Non-inferiority Study - SATISFACTION
Brief Title: Efficacy and Safety of mAnnitol in Bowel Preparation During Elective Colonoscopy and Comparison With Moviprep®
Acronym: SATISFACTION
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NTC srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Mannitol_03-2018; 2019-002856-18 (EudraCT Number)
Record Dates: First submitted 2020-11-30; First posted 2021-02-18 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Elective Colonoscopy
Keywords: Colonoscopy preparation; Bowel cleansing; Gas; Mannitol
MeSH Terms: conditions — Mucopolysaccharidosis IV | interventions — MoviPrep

STUDY DESIGN:
Intervention Model Description: A randomized, parallel-group study.
Who Masked: Outcomes Assessor
Masking Description: Endoscopist-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase II: NTC015 low dose (Mannitol 50 g) (Experimental): One day single dose preparation same day of colonoscopy
  Interventions: Drug: Phase II: NTC015 low dose
- Phase II: NTC015 medium dose (Mannitol 100 g) (Experimental): One day single dose preparation same day of colonoscopy
  Interventions: Drug: Phase II: NTC015 medium dose
- Phase II: NTC015 high dose (Mannitol 150 g) (Experimental): One day single dose preparation same day of colonoscopy
  Interventions: Drug: Phase II: NTC015 high dose
- Phase III: NTC015 selected dose (Experimental): One day single dose preparation same day of colonoscopy
  Interventions: Drug: Phase III: NTC015 selected dose
- Phase III: Polyethylene glycol plus ascorbate solution (2L PEG ASC) (Moviprep®) (Active Comparator): Two litres of Moviprep® taken according to split-dose regimen (to commence in the evening before colonoscopy)
  Interventions: Drug: Phase III: Polyethylene glycol plus ascorbate solution (2L PEG ASC)

INTERVENTIONS:
Drug: Phase II: NTC015 low dose — Participants should self administer the preparation within 30 minutes and drink clear liquid according to local practice at the centre to prevent dehydration
  Arms: Phase II: NTC015 low dose (Mannitol 50 g)
Drug: Phase II: NTC015 medium dose — Participants should self administer the preparation within 30 minutes and drink clear liquid according to local practice at the centre to prevent dehydration
  Arms: Phase II: NTC015 medium dose (Mannitol 100 g)
Drug: Phase II: NTC015 high dose — Participants should self administer the preparation within 60 minutes and drink clear liquid according to local practice at the centre to prevent dehydration
  Arms: Phase II: NTC015 high dose (Mannitol 150 g)
Drug: Phase III: NTC015 selected dose — Participants should self administer the preparation within 30 minutes and drink clear liquid according to local practice at the centre to prevent dehydration
  Arms: Phase III: NTC015 selected dose
Drug: Phase III: Polyethylene glycol plus ascorbate solution (2L PEG ASC) — The instructions for product administration are followed according to the Summary of Product Characteristics.
  One treatment consists of two litres of Moviprep® taken according to split-dose regimen.
  The first litre of Moviprep® is prepared by dissolving one sachet A and one sachet B together in water to make one litre of solution. The reconstituted solution must be drunk over a period of one to two hours the evening before colonoscopy. About half a litre of clear liquid should be drunk in the next hour to prevent dehydration according to local practice at the centre. This process should be repeated with a second litre of Moviprep® prepared by dissolving one sachet A and one sachet B together in water to make one litre of solution in the early morning of the day of the procedure.
  Other Names: Moviprep®
  Arms: Phase III: Polyethylene glycol plus ascorbate solution (2L PEG ASC) (Moviprep®)

SUMMARY:
The purpose of this dose finding/comparative efficacy study is to first single out the most appropriate dose of mannitol for bowel preparation (phase II) and, subsequently, demonstrate the non-inferiority of the efficacy of single dose mannitol vs standard split 2L PEG ASC (Moviprep®) (phase III) in bowel preparation for colonoscopy .

DETAILED DESCRIPTION:
Study Start and Study Completion dates relative to the Phase II/III are reported here:

Phase II (Patients n. 183)

* Date of first enrolment: 18 June 2020
* Date LPLV: 12 November 2020

Phase III (Patients n. 703)

* Date of first enrolment: 2 March 2021
* Date LPLV: 16 July 2021

Date on which the study was entered in the EudraCT database: 13 October 2020

ELIGIBILITY:
Inclusion Criteria:

1. Ability of patient to consent and provide signed written informed consent
2. Age ≥ 18 years
3. Males and females scheduled for elective (screening, surveillance or diagnostic) colonoscopy to be prepared and performed according to the European Society of Gastrointestinal Endoscopy (ESGE) Guideline
4. Patients willing and able to complete the entire study and to comply with instructions

Exclusion Criteria:

1. Pregnancy or breastfeeding. Females of childbearing potential must have a negative pregnancy test at Visit 2 and must practice one of the following methods of birth control throughout the study period (unless postmenopausal or surgically sterile, or whose sole sexual partner has had a successful vasectomy): oral, implantable, or injectable contraceptives (for a minimum of three months before study entry) in combination with a condom; intrauterine device in combination with a condom; double barrier method (condom and occlusive cap with spermicidal foam/gel/film/cream/suppository).
2. Severe renal failure: glomerular filtration rate (eGFR) < 30 ml/min/1.73 m2 estimated by means of simplified MDRD equation.
3. Severe heart failure: NYHA Class III-IV.
4. Severe anaemia (Hb ≤ 8 g/dl).
5. Severe acute and chronically active Inflammatory Bowel Disease; patients in clinical remission (Crohn's Disease Activity Index - CDAI < 150 for Crohn Disease and Partial Mayo Score ≤ 2 for Ulcerative Colitis) are allowed.
6. Chronic liver disease Child-Pugh class B or C.
7. Electrolyte disturbances (Na, Cl, K, Ca or P out of normal ranges).
8. Recent (< 6 months) symptomatic acute ischemic heart disease.
9. History of significant gastrointestinal surgeries, including colon resection, sub-total colectomy, abdominoperineal resection, de-functioning colostomy or ileostomy, Hartmann's procedure and other surgeries involving the structure and function of the colon.
10. Use of laxatives, colon motility altering drugs and/or other substances (e.g. simethicone) that can affect bowel cleansing or visibility during colonoscopy within 24 hours prior to colonoscopy.
11. Suspected bowel obstruction or perforation.
12. Indication for partial colonoscopy.
13. Patients who have received an investigational drug or therapy within 5 half-lives of the first visit.
14. Patients previously screened for participation in this study.
15. Hypersensitivity to the active ingredients or to any of the excipients of the study drugs.
16. Contraindication to Moviprep® (only for phase III).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 886 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianpiero Manes, Dr., Principal Investigator — ASST Rhodense - Presidi di Rho e Garbagnate
Locations (35):
- France (4):
  - Centre Hospitalier Henri Duffaut, Avignon
  - Hospices civils de Lyon, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
- Germany (4):
  - Klinikum der Stadt Ludwigshafen, Ludwigshafen
  - Praxis für Gastroenterologie und Fachärztliche Innere Medizin, Im Haus der Gesundheit, Ludwigshafen am Rhein
  - Katholisches Klinikum Mainz, Mainz
  - Klinikum Worms Medizinische Klinik II, Worms
- Italy (19):
  - IRCCS "Saverio De Bellis", Castellana Grotte, BA
  - Fondazione Poliambulanza - Istituto Ospedaliero, Brescia, BR
  - ASSL Carbonia - Presidio Ospedaliero CTO di Iglesias, Iglesias, CI
  - Ospedale Valduce, Como, CO
  - Fondazione Casa Sollievo Della Sofferenza, San Giovanni Rotondo, FG
  - ASST Rhodense - Presidi di Rho e Garbagnate, Garbagnate Milanese, MI
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico di Milano, Milan, MI
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - IRCCS Ospedale San Raffaele, Milan, MI
  - Istituto Europeo di Oncologia, Milan, MI
  - IRCCS Policlinico San Donato, San Donato Milanese, MI
  - Azienda USL di Modena - Ospedale Ramazzini di Carpi, Carpi, MO
  - Azienda Ospedaliero Universitaria Pisana- Ospedale Cisanello, Pisa, PI
  - Centro di Riferimento Oncologico IRCCS, Aviano, PN
  - Policlinico Universitario A. Gemelli, Roma, RO
  - Presidio Ospedaliero Santa Chiara, Trento, TN
  - Ospedale Sacro Cuore, Negrar, VR
  - Azienda Ospedaliero-Universitaria Maggiore della Carità, Novara
  - ASST Sette Laghi - Ospedale di Circolo e Fondazione Macchi, Varese
- Russia (8):
  - Irkutsk State Medical Academy of Postgraduate Education, Irkutsk
  - Clinical Hospital of Russian Railways N.A. Semashko, Moscow
  - Moscow Clinical Research and Practical Center of the Department of Health, Moscow
  - State Central Clinical Hospital A. N. Ryzhykh, Moscow
  - Railway Clinical Hospital, Rostov
  - Private educational organization of higher education "Medical University "Reaviz", Samara
  - Medical Center of Diagnostics and Prevention, Yaroslavl
  - Regional Oncological Clinical Hospital, Yaroslavl

REFERENCES:
- [Derived] Tontini GE, Spada C, Uebel P, Cannizzaro R, Ciprandi G, Vecchi M. Assessment of Patient-Reported Outcome Measures in Patients Undergoing Bowel Preparation With Mannitol for Colonoscopy: The SATISFACTION Study. JGH Open. 2025 Aug 7;9(8):e70237. doi: 10.1002/jgh3.70237. eCollection 2025 Aug. PMID 40786127
- [Derived] Carnovali M, Spada C, Uebel P, Bocus P, Cannizzaro R, Cavallaro F, Cesana BM, Cesaro P, Costamagna G, Di Paolo D, Ferrari AP, Hinkel C, Kashin S, Massella A, Melnikova E, Orsatti A, Ponchon T, Prada A, Radaelli F, Sferrazza S, Soru P, Testoni PA, Tontini GE, Vecchi M, Fiori G; SATISFACTION Study Group. Factors influencing the presence of potentially explosive gases during colonoscopy: Results of the SATISFACTION study. Clin Transl Sci. 2023 May;16(5):759-769. doi: 10.1111/cts.13486. Epub 2023 Feb 17. PMID 36799346

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study period:
  * Phase II study initiation date: 22 June 2020
  * Phase II LPLV: 12 November 2020
  * Phase III study initiation date: 2 March 2021
  * Phase III LPLV: 16 July 2021
  * Phase II: 6 centres in Italy, 2 centres in Germany and 1 centre in France
  * Phase III: 32 centres located in Italy, Germany, France, and Russia
Pre-assignment Details: Phase II Planned sample size n.150; screened patients n.199; screen failures n.16; randomized patients n.183; completed patients: 179
  Phase III Planned sample size n.696; screened patients n. 841; withdrawal patients n. 7; screen failures n. 131; randomized patients n.703; completed patients: 683
Groups:
- Phase II: NTC015 Low Dose: Mannitol 50 g administered as single dose
- Phase II: NTC015 Medium Dose: Mannitol 100 g administered as single dose
- Phase II: NTC015 High Dose: Mannitol 150 g administered as single dose
- Phase III: NTC015 Selected Dose: Mannitol 100 g selected from phase II, single dose
- Phase III: 2L PEG ASC (Moviprep®): 2 L polyethylene glycol plus ascorbate solution, split-dose regimen
Period: Overall Study
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose | Phase III: NTC015 Selected Dose | Phase III: 2L PEG ASC (Moviprep®)
Started | 66 | 57 | 60 | 352 | 351
Completed | 65 | 57 | 57 | 338 | 345
Not Completed | 1 | 0 | 3 | 14 | 6
Not completed — Other | 1 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 9 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Set
Groups:
- Phase III: 2L PEG ASC (Moviprep®): 2 L polyethylene glycol plus ascorbate solution, split dose
- Total: Total of all reporting groups
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose | Phase III: NTC015 Selected Dose | Phase III: 2L PEG ASC (Moviprep®) | Total
Number analyzed (Participants) | 66 | 57 | 60 | 352 | 351 | 886
Age, Customized [Mean (Standard Deviation); unit: years]
  Age at study entry | 57.55 (11.15) | 54.4 (11.19) | 53.8 (13.78) | 54.8 (12.65) | 54.6 (12.71) | 54.7 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 36 | 219 | 196 | 513
  Male | 36 | 25 | 24 | 133 | 155 | 373
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 3 | 4 | 4 | 13
  Not Hispanic or Latino | 63 | 54 | 56 | 343 | 344 | 860
  Unknown or Not Reported | 1 | 3 | 1 | 5 | 3 | 13
Female reproductive status [Count of Participants; unit: Participants] — Population: Percentages were computed on female patients belonging to the PP Population.
  Participants
    number analyzed (Participants) | 30 | 32 | 36 | 219 | 196 | 513
    Childbearing potential | 8 | 6 | 15 | 103 | 100 | 232
    Menopause | 20 | 23 | 21 | 106 | 87 | 257
    Sterile | 2 | 3 | 0 | 9 | 8 | 22
    Other | 0 | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase II - Dose Finding: Proportion of Patients With Adequate Bowel Cleansing
Description: Proportion of patients with adequate bowel cleansing, defined as BBPS total score ≥ 6, with a score for each of the three colon segments ≥ 2 during colonoscopy after standard washing and air insufflation for luminal distension.
  The mannitol dose to be used in phase III was singled out on an algorithm that calculated a total score for each dose starting from the scores assigned to the three main criteria through a ranking system and proportionally to the importance given to each main criterion: A - rate of adequate bowel cleansing (most important - primary endpoint), B - rate of patients in safe conditions and C - clinical judgement score (least important - partially based on subjective assessments).
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed
Population: Percentages were computed on patients belonging to the PP population.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Groups:
- Phase II: NTC015 Low Dose: Mannitol 50 g administered as a single dose
- Phase II: NTC015 Medium Dose: Mannitol 100 g administered as a single dose
- Phase II: NTC015 High Dose: Mannitol 150 g administered as a single dose
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose
Number analyzed (Participants) | 60 | 54 | 49
Proportion of patients | 0.75 [0.64 to 0.86] | 0.94 [0.88 to 1] | 0.94 [0.87 to 1]

2. Primary Outcome: Phase III - Non-inferiority: Proportion of Patients With Adequate Bowel Cleansing
Description: Proportion of patients with adequate bowel cleansing, defined as BBPS total score ≥ 6, with a score for each of the three colon segments (right; transverse, including flexures; and left, including sigmoid and rectum) ≥ 2 during colonoscopy after standard washing and air insufflation for luminal distension.
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed, at least 4 hours after end of intake, following product instruction as per protocol
Population: Percentages were computed on patients belonging to the PP Population.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Groups:
- Phase III: NTC015 Selected Dose: Mannitol 100 g selected in phase II, single dose
- Phase III: 2 L PEG ASC (Moviprep®): 2 L polyethylene glycol plus ascorbate solution, split dose
Arm/Group | Phase III: NTC015 Selected Dose | Phase III: 2 L PEG ASC (Moviprep®)
Number analyzed (Participants) | 325 | 332
Proportion of patients | 0.91 [0.88 to 0.94] | 0.95 [0.93 to 0.98]

3. Secondary Outcome: Phase II - Dose Finding: Caecal Intubation Rate
Description: The percentage of patients with appendiceal orifice visible to the endoscopist. Evaluation will be performed during conduction of colonoscopy run on visit 4. Timing for treatment administration was described in the protocol and change among arms.
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed
Population: Percentages were computed on patients belonging to the PP population.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose
Number analyzed (Participants) | 60 | 54 | 49
Proportion of patients | 0.92 [0.85 to 0.99] | 1 [1 to 1] | 1 [1 to 1]

4. Secondary Outcome: Phase II - Dose Finding: Adherence to Bowel Preparation
Description: Proportion of patient that completely taken assigned mannitol dose.
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed, 4 hours after the end of study drug self-administration, before colonoscopy
Population: Percentages were computed on patients belonging to the PP population. Overall Number of Participants Analyzed referred to patient that completely taken assigned mannitol dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose
Number analyzed (Participants) | 60 | 54 | 49
Participants | 60 | 54 | 49

5. Secondary Outcome: Phase II - Dose Finding: Ease of Use
Description: Descriptive statistics (Mean) of Numeric Rating Scale (NRS) values ranging from 0 (very difficult) to 10 (very easy).
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed. 4 hours after the end of study drug self-administration, before colonoscopy (please refer to protocol)
Population: Percentages were computed on patients belonging to the PP population.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose
Number analyzed (Participants) | 60 | 54 | 49
Score | 9.6 (0.70) | 9.3 (1.09) | 9.1 (1.36)

6. Secondary Outcome: Phase II - Dose Finding: Willingness to Reuse the Preparation
Description: Proportion of patient who confirmed that they would like to reuse the preparation for other colonoscopies.
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed. 4 hours after the end of study drug self-administration, before colonoscopy
Population: Percentages were computed on patients belonging to the PP population.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose
Number analyzed (Participants) | 60 | 54 | 49
Participants
  Yes | 60 | 51 | 46
  No | 0 | 3 | 3

7. Secondary Outcome: Phase II - Dose Finding: Treatment Acceptability
Description: Descriptive statistics (Mean) of Numeric Rating Scale (NRS) values ranging from 0 (terrible) to 10 (very good).
Time Frame: as for outcome 6
Population: Percentages were computed on patients belonging to the PP population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose
Number analyzed (Participants) | 60 | 54 | 49
score on a scale | 9.2 (1.01) | 8.3 (1.49) | 8.0 (1.94)

8. Secondary Outcome: Phase II - Pharmacokinetic Parameter: Peak Plasma Concentration
Description: descriptive statistics (mean) of peak plasma concentration (Cmax) as pharmacokinetic parameter.
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed. Before mannitol self-administration and 8 hours (T8) after completion of mannitol self-administration
Population: Percentages were computed on patients belonging to the PK population.
Measure: Mean (Standard Deviation); unit: Mannitol plasma concentrations (mg/mL)
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose
Number analyzed (Participants) | 15 | 11 | 17
Mannitol plasma concentrations (mg/mL) | 0.6304 (0.14536) | 1.0236 (0.27877) | 1.3729 (0.38338)

9. Secondary Outcome: Phase II - Pharmacokinetic Parameter: Time to Maximum Concentration
Description: Descriptive statistics (Median) of time to maximum concentration (tmax) as pharmacokinetic parameter.
Time Frame: as for outcome 8
Population: Percentages were computed on patients belonging to the PK population.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose
Number analyzed (Participants) | 15 | 11 | 17
Hours | 1.1173 (0.36110) | 1.3636 (0.52259) | 1.4488 (0.80422)

10. Secondary Outcome: Phase II - Pharmacokinetic Parameter: Area Under the Curve
Description: Descriptive statistics (Mean) of area under the curve from t0 to the last blood sampling time point (AUC 0-t8), as pharmacokinetic parameter.
Time Frame: as for outcome 8
Population: Percentages were computed on patients belonging to the PK population.
Measure: Mean (Standard Deviation); unit: mg/mL*hours
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose
Number analyzed (Participants) | 15 | 11 | 17
mg/mL*hours | 2.2313 (0.52086) | 4.1591 (1.34820) | 5.8476 (2.36432)

11. Secondary Outcome: Phase II - Pharmacokinetic Parameter: Terminal Elimination Half Life
Description: Descriptive statistics (Mean) of elimination half life (t1/2), as pharmacokinetic parameter.
Time Frame: as for outcome 8
Population: Percentages were computed on patients belonging to the PK population.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose
Number analyzed (Participants) | 13 | 7 | 11
Hours | 2.5838 (0.83985) | 2.4186 (0.57883) | 2.6782 (0.48912)

12. Secondary Outcome: Phase III - Non-inferiority: Adenoma Detection Rate
Description: The percentage of patients with at least one lesion detected.
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed
Population: Percentages were computed on patients belonging to the Full Analysis Set.
Measure: Number; unit: Number of patients
Arm/Group | Phase III: NTC015 Selected Dose | Phase III: 2L PEG ASC (Moviprep®)
Number analyzed (Participants) | 333 | 347
Number of patients
  Adenoma detection rate - Yes | 98 | 103
  Adenoma detection rate - No | 235 | 244

13. Secondary Outcome: Phase III - Non-inferiority: Ottawa Bowel Preparation Scale (OBPS)
Description: Ottawa scale is used to measure the quality of the preparation in three different parts of the colon before washing and insufflation. descriptive statistics (Mean) of the total score (from 0 excellent to 14 inadequate).
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed
Population: Percentages were computed on patients belonging to the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase III: NTC015 Selected Dose | Phase III: 2L PEG ASC (Moviprep®)
Number analyzed (Participants) | 332 | 347
score on a scale | 4.4 (3.08) | 3.6 (2.52)

14. Secondary Outcome: Phase III - Non-inferiority: Caecal Intubation Rate
Description: The percentage of patients with appendiceal orifice visible to the endoscopist.
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed
Population: Percentages were computed on patients belonging to the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase III: NTC015 Selected Dose | Phase III: 2L PEG ASC (Moviprep®)
Number analyzed (Participants) | 333 | 347
Participants
  Yes | 327 | 345
  No | 6 | 2

15. Secondary Outcome: Phase III - Non-inferiority: Bowel Cleansing Impact Review (BOCLIR) (Italian Sites Only)
Description: The BOCLIR is a questionnaire filled in by patients to measure the acceptability and tolerability of bowel cleansers consisting of three unidimensional scales (satisfaction, symptoms and activity limitations) with good psychometric and scaling properties. Item responses are summed to provide a score for each scale and a total score. The satisfaction scale contains eight items and the score ranges from 0 (highly satisfied) to 32 (highly dissatisfied). The symptoms scale includes 14 items and the score ranges from 0 (no symptoms) to 42 (severe symptoms).
  The activity limitations scale is made up of 12 items and the score ranges from 0 (no effect on activities) to 36 (activities greatly affected). The total score is the sum of the three scales and ranges from 0 to 110. Patients who report a worse experience in terms of the three factors score higher on the BOCLIR scale.
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed. After the end of study drug self-administration, before colonoscopy
Population: Percentages were computed on patients belonging to Italian centers in the Safety set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase III: NTC015 Selected Dose | Phase III: 2L PEG ASC (Moviprep®)
Number analyzed (Participants) | 236 | 240
score on a scale | 23.5 (13.48) | 31.5 (16.26)

16. Secondary Outcome: Phase III - Non-inferiority: Adherence to Bowel Preparation With Mannitol and With Moviprep®.
Description: Proportion of patients that completely taken, partially taken or not taken assigned mannitol dose
Time Frame: as for outcome 6
Population: Percentages were computed on patients belonging to the Safety set who have been administered questionnaire on adherence and acceptability.
Measure: Number; unit: Number of patients
Arm/Group | Phase III: NTC015 Selected Dose | Phase III: 2L PEG ASC (Moviprep®)
Number analyzed (Participants) | 341 | 347
Number of patients
  Completely taken (fully drinked) | 341 | 341
  Partially taken | 0 | 6

17. Secondary Outcome: Phase III - Non-inferiority: Ease of Use
Description: Descriptive statistics (Mean) of Numeric Rating Scale (NRS) values ranging from 0 (very difficult) to 10 (very easy).
Time Frame: as for outcome 6
Population: Percentages were computed on patients belonging to the Safety set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase III: NTC015 Selected Dose | Phase III: 2L PEG ASC (Moviprep®)
Number analyzed (Participants) | 341 | 347
score on a scale | 9.3 (1.41) | 8.5 (2.00)

18. Secondary Outcome: Phase III - Non-inferiority: Willingness to Reuse the Preparation
Description: Proportion of patient who confirmed that they would like to reuse the preparation for other colonoscopies.
Time Frame: as for outcome 6
Population: Percentages were computed on patients belonging to the Safety set who have been administered questionnaire on adherence and ac ceptability.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase III: NTC015 Selected Dose | Phase III: 2L PEG ASC (Moviprep®)
Number analyzed (Participants) | 341 | 347
Participants
  Yes | 331 | 272
  No | 10 | 75

19. Secondary Outcome: Phase III - Non-inferiority: Treatment Acceptability
Description: Descriptive statistics (Mean) of Numeric Rating Scale (NRS) values ranging from 0 (terrible) to 10 (very good).
Time Frame: as for outcome 6
Population: Percentages were computed on patients belonging to the Safety set.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Phase III: NTC015 Selected Dose: Mannitol 100g selected in phase II, single dose
Arm/Group | Phase III: NTC015 Selected Dose | Phase III: 2L PEG ASC (Moviprep®)
Number analyzed (Participants) | 341 | 347
score on a scale | 8.3 (1.74) | 5.6 (2.67)

20. Other Pre Specified Outcome: Phase II - Dose Finding: Patients in Safe Condition Related to Potentially Critical Concentrations of Gases (H2/CH4)
Description: Proportion of patients in safe condition for intestinal gases defined as concentration of potentially critical concentrations of gases (H2>4% and CH4 >5%)
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed after standard washing and air insufflation for luminal distension
Population: Percentages were computed on patients belonging to the PP population evaluable for potentially dangerous levels of H2 and CH4
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose
Number analyzed (Participants) | 60 | 54 | 49
Participants
  Proportion of patients with potentially dangerous levels of H2 | 0 | 0 | 0
  Proportion of patients with potentially dangerous levels of CH4 | 0 | 0 | 0

21. Other Pre Specified Outcome: Phase II - Dose Finding: Incidence of Adverse Events
Description: Incidence of adverse events occuring starting from enrollment
Time Frame: Visit 2 (≤ 7 days before Visit 4), Visit 3 (≤ 7 days before Visit 4) and Visit 4 (during the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed)
Population: Percentages were computed on patients belonging to the Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose
Number analyzed (Participants) | 65 | 57 | 57
Participants
  Patients with at least one TEAE | 7 | 11 | 19
  Patients with at least one TESAE | 0 | 0 | 1
  Patients with at least one TEAE related to study drug | 2 | 6 | 12
  Patients with at least one TESAE related to study drug | 0 | 0 | 0
  Patients with at least one TESAE related to colonoscopy | 0 | 0 | 0
  Patients with at least one TEAE related to colonoscopy | 1 | 1 | 2
  Patients with at least one TEAE leading to study drug withdrawal | 0 | 0 | 1
  Patients with at least one TESAE leading to colonoscopy interruption | 0 | 0 | 0
  Patients with at least one fatal TESAE | 0 | 0 | 0
  Patients with at least one AESI | 1 | 7 | 11

22. Other Pre Specified Outcome: Phase II - Dose Finding: Proportion of Patients With Clinically Significant Change of Haematological and Chemical Parameters From Baseline
Description: Proportion of patients with change from baseline considered clinically significant by the Investigator of haematological and chemical parameters (CBC, creatinine, BUN, eGFR, ALT, AST, glucose, electrolytes) 4 hours and 8 hours after completion of study drug self-administration.
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed. 4 hours and 8 hours after completion of study drug self administration
Population: Percentages were computed on patients belonging to the Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose
Number analyzed (Participants) | 65 | 57 | 57
Participants
  Patients with at least one clinically significant abnormality (hematological parameters) | 0 | 0 | 2
  Patients with at least one clinically significant abnormality (chemical parameters) | 1 | 0 | 2

23. Other Pre Specified Outcome: Phase II - Dose Finding: Proportion of Patients With Clinically Significant Change of Vital Signs During Colonoscopy
Description: Proportion of patients with change of vital signs during colonoscopy considered clinically significant by the Investigator (heart rate and pulse oximetry).
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose
Number analyzed (Participants) | 65 | 57 | 57
Participants | 0 | 0 | 0

24. Other Pre Specified Outcome: Phase III - Dose Finding:Patients in Safe Condition Related to Potentially Critical Concentration of Gases (H2/CH4)
Description: Proportion of patients in safe condition for intestinal gases defined as concentration of potentially critical concentration of gases (H2>4% and CH4 >5%)
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed
Population: Percentages were computed on patients belonging to the safety set evaluable for potentially dangerous levels of H2 and CH4. Some patients were excluded from the analysis because their gas concentrations were measured through a device with malfunction issues
Measure: Count of Participants; unit: Participants
Groups:
- Phase III: 2L PEG ASC (Moviprep®): 2 L polyethylene glycol plus ascorbate solution
Arm/Group | Phase III: NTC015 Selected Dose | Phase III: 2L PEG ASC (Moviprep®)
Number analyzed (Participants) | 331 | 342
Participants
  Proportion of patients with potentually dangerous levels H2 | 0 | 0
  Proportion of patients with potentually dangerous levels CH4 | 0 | 0

25. Other Pre Specified Outcome: Phase III - Non-inferiority: Incidence of Adverse Events
Description: Incidence of adverse events occuring starting from enrollment
Time Frame: as for outcome 21
Population: Percentages were computed on patients belonging to the Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase III: NTC015 Selected Dose | Phase III: 2L PEG ASC (Moviprep®)
Number analyzed (Participants) | 343 | 347
Participants
  Patients with at least one TEAE | 52 | 36
  Patients with at least one TESAE | 3 | 0
  Patients with at least one TEAE related to study drug | 32 | 14
  Patients with at least one TESAE related to study drug | 3 | 0
  Patients with at least one TEAE related to study drug leading to study drug withdrawal | 1 | 1
  Patients with at least one TESAE related to study drug leading to study drug withdrawal | 0 | 0
  Patients with at least one TEAE related to colonoscopy | 5 | 2
  Patients with at least one TESAE related to colonoscopy | 0 | 0
  Patients with at least one TEAE leading to study drug withdrawal | 1 | 1
  Patients with at least one TEAE leading to colonoscopy interruption | 1 | 1
  Patients with at least one fatal TESAE | 0 | 0
  Patients with at least one treatment-emergent AESI | 27 | 9

26. Other Pre Specified Outcome: Phase III - Non-inferiority: Proportion of Patients With Clinically Significant Change of Haematological and Chemical Parameters From Baseline
Description: as for outcome 22
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed. 4 hours and 8 hours after completion of study drug self-administration
Population: Percentages were computed on patients belonging to the Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase III: NTC015 Selected Dose | Phase III: 2L PEG ASC (Moviprep®)
Number analyzed (Participants) | 343 | 347
Participants
  Patients with at least one clinically significant abnormality (Hematology) | 2 | 0
  Patients with at least one clinically significant abnormality (Clinical chemistry) | 12 | 5

27. Other Pre Specified Outcome: Phase III - Non-inferiority: Proportion of Patients With Change of Vital Signs From Baseline and During Colonoscopy
Description: Proportion of patients with change of vital signs from baseline considered clinically significant by the Investigator (heart rate, systolic and diastolic blood pressure), as well as clinically significant change during colonoscopy of pulse oximetry, systolic and diastolic blood pressure and heart rate.
Time Frame: During the colonoscopy procedure, carried out within 7 days of the screening visit, the evaluation is performed, prior to colonoscopy
Population: Percentages were computed on patients belonging to the Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase III: NTC015 Selected Dose | Phase III: 2L PEG ASC (Moviprep®)
Number analyzed (Participants) | 343 | 347
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Phase II and III: Adverse events where monitored during 4 visits of the study: from signature of the informed consent form up to and including the day of colonoscopy, up to 4 weeks (i.e., day in which patient performed the last assessment planned in the study protocol and thus complete the study). After the drug intake adverse event was checked during day of colonoscopy. In case of serious adverse event the clinical situation was monitored until resolution
Groups:
- Phase III: NTC015 Selected Dose: Mannitol 100g selected from phae II, single dose
- Phase III:2 L PEG ASC (Moviprep®): 2 L polyethylene glycol plus ascorbate solution, split dose
Arm/Group | Phase II: NTC015 Low Dose | Phase II: NTC015 Medium Dose | Phase II: NTC015 High Dose | Phase III: NTC015 Selected Dose | Phase III:2 L PEG ASC (Moviprep®)
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/57 | 0/57 | 0/343 | 0/347
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/57 | 1/57 | 3/343 | 0/347
Other Adverse Events (participants affected / at risk) | 3/65 | 8/57 | 17/57 | 25/343 | 9/347
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase II: NTC015 Low Dose (N=65) | Phase II: NTC015 Medium Dose (N=57) | Phase II: NTC015 High Dose (N=57) | Phase III: NTC015 Selected Dose (N=343) | Phase III:2 L PEG ASC (Moviprep®) (N=347)
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II: NTC015 Low Dose (N=65) | Phase II: NTC015 Medium Dose (N=57) | Phase II: NTC015 High Dose (N=57) | Phase III: NTC015 Selected Dose (N=343) | Phase III:2 L PEG ASC (Moviprep®) (N=347)
diverticulum intestinal (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 8 (8) | 15 (15) | 2 (2)
large intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (3) | 10 (10) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT04759885/Prot_SAP_000.pdf